CLINICAL TRIAL: NCT06723522
Title: The Efficacy and Brain Mechanism of High Definition Transcranial Direct Current Stimulation of Right Inferior Frontal Gyrus to Improve Social Impairments in Children with Autism Spectrum Disorder: a Randomized, Double-blind, Controlled Study
Brief Title: High Definition Transcranial Direct Current Stimulation of Right Inferior Frontal Gyrus to Improve Social Impairments in Children with Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Xuerong Luo, Doctor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYEC2024-0306
Record Dates: First submitted 2024-11-28; First posted 2024-12-09 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: autism; tDCS; social; fNIRS; RCT
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): Received a dose of 2 mA HD-tDCS stimulation lasted for 20 min, with 30 s of ramp-up and ramp-down before and after the 20-min stimulation, respectively.
  Interventions: Device: HD-tDCS
- Sham group (Sham Comparator): Received 1 min of ramping up/down without experiencing 2 mA HD-tDCS stimulation lasted for 20 min.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: HD-tDCS — 2 mA HD-tDCS of right inferior frontal gyrus lasting for 10 days, each stimulation lasted for 20 min, with 30 s of ramp-up and ramp-down before and after the 20-min stimulation, respectively.
  Arms: Active group
Device: Sham (No Treatment) — Received 1 min of ramping up/down without experiencing 2 mA HD-tDCS stimulation lasted for 20 min.
  Arms: Sham group

SUMMARY:
The goal of this clinical trial is to learn if high definition transcranial direct current stimulation (HD-tDCS) of right inferior frontal gyrus works to improve social impairments in children with autism spectrum disorder (ASD). It will also learn about the underlying brain mechanism. The main questions it aims to answer are:

* Does HD-tDCS of right inferior frontal gyrus improve social impairments in children with ASD?
* What are the underlying brain mechanisms by which the HD-tDCS of right inferior frontal gyrus improves social impairments in children with ASD? Researchers will compare participants received active HD-tDCS to controls received sham HD-tDCS (performed to mimic the sensation induced by real HD-tDCS before and after the stimulation) to see if HD-tDCS of right inferior frontal gyrus improves social impairments in children with ASD.

Participants will:

* Receive a dose of 2 mA HD-tDCS of right inferior frontal gyrus lasting for 10 days.
* Receive social functioning assessment, functional near-infrared spectroscopy and electroencephalography measurement before and after stimulation
* Visit the clinic once every 2 weeks for checkups and tests, a total of 2 times.

ELIGIBILITY:
Inclusion Criteria:

* had to be 3-18 years old; be diagnosed with ASD (according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and Autism Diagnostic Interview - Revised (ADI-R).

Exclusion Criteria:

* with other comorbid neuropsychiatric conditions (i.e., schizophrenia spectrum disorders and mood disorders) or neurological disorders (i.e., head trauma and epilepsy).

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Social function as measured by the Social Responsiveness Scale-2nd Edition(SRS-2) | Social functioning was assessed before stimulus onset, immediately after stimulus completion, at week 2 after completion, and at week 4 after completion.
  SRS-2 is a highly reliable and sensitive scale to measure social function in RCTs involving individuals with autism.

SECONDARY OUTCOMES:
The resting-state functional connectivity between the right inferior frontal gyrus and other brain regions involving social function as measured by functional near-infrared spectroscopy | before stimulus onset, immediately after stimulus completion, at week 2 after completion, and at week 4 after completion.
  Functional changes in individuals with autism have been found to be associated with social impairment in these individuals. Functional near-infrared spectroscopy (fNIRS) is a non-invasive, portable and body-motion tolerant neuroimaging technique that has been used to measure changes in functional connectivity between different brain networks.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No